CLINICAL TRIAL: NCT01215682
Title: Vitamin D Supplementation, Upper Respiratory Tract Infections, Immune and Physical Functions in Adolescent Swimmers
Brief Title: Vitamin D Supplementation and Upper Respiratory Tract Infections in Adolescent Swimmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Gal Raz-Dubnov MD, MSc, senior physician, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SHEBA-10-7762-GDR-CTIL
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Upper Respiratory Tract Infections
Keywords: infections; immune system; vitamin D; sport; children
MeSH Terms: conditions — Respiratory Tract Infections; Infections | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vit D (Active Comparator)
  Interventions: Dietary Supplement: vitamin D
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: vitamin D — 2000 IU/day of vitamin D3 as a once-daily dose
  Arms: vit D
Dietary Supplement: placebo — sweetened water
  Arms: placebo

SUMMARY:
Background: The medical and economic burden of upper respiratory tract infections (URTIs) is extremely high, while prevention and treatment options are limited. Therefore, there is a constant need for new methods in order to significantly decrease such morbidity. Extensive evidence shows that vitamin D is associated with respiratory health, including in the prevention and treatment of URTIs. Competitive swimmers have a high prevalence of URTIs, and can serve as a model for research in this field.

The study hypothesis is that vitamin D supplementation to young swimmers with low vitamin D levels will reduce the frequency, length, and severity of URTIs and their accompanying functional impairment, while improving cellular immune function and physical function.

Methods: After screening 100 competitive adolescent swimmers to obtain ~60 with low serum levels of vitamin D, this study group will be randomized to receive either vitamin D supplementation (2000 IU/d) or placebo, given in a double blinded fashion for three months. Participants will fill a daily questionnaire regarding frequency, length and severity of URTIs symptoms and functional impairment. Blood will be drawn to evaluate changes in vitamin D status (25(OH)D) and immune function among study participants at the beginning of the study and after supplementation. Physical function on land and in water will also be assessed.

Expected results: Increase in serum 25(OH)D levels following supplementation will significantly decrease the frequency, length and severity of URTI's and their functional impairment, while enhancing the cellular immune system function and physical capacity.

ELIGIBILITY:
Inclusion Criteria:

* members of swimming team
* training at least 15 hours/week
* low vitamin D plasma levels (<30 ng/ml)
* signed consent forms

Exclusion Criteria:

* chronic health conditions
* taking prescription medications
* taking diet supplementations

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
URI frequency | 3 months
  URI frequency will be measured in both groups, starting 4 weeks after initiating the suplementation. Analysis will also assess differences by sex or initial vitamin D levels, as well as by immune function changes.
URI duration | 3 months
  URI duration will be measured in both groups, starting 4 weeks after initiating the suplementation. Analysis will also assess differences by sex or initial vitamin D levels, as well as by immune function changes.
UTI severity | 3 months
  URI severity will be measured in both groups, starting 4 weeks after initiating the suplementation. Analysis will also assess differences by sex or initial vitamin D levels, as well as by immune function changes.

SECONDARY OUTCOMES:
plasma vitamin D levels | 3 months
immune system function | 3 months
  T-cell receptor excision circles (TREC), T cell receptor repertoire, B-cell receptor excision circles (BREC). Comparison will be made with changes in vitamin D levels and with URI characteristics.
physical function | 3 months
  absence from school or training, land and swimming fitness tests. Comparison will be made with changes in vitamin D levels.

CONTACTS AND LOCATIONS:
Overall Officials: Gal Dubnov-Raz, MD MSc, Principal Investigator — Sheba Medical Center; Naama W Constantini, MD, Principal Investigator — Hadassah Medical Organziation; Avner Cohen, MD, Principal Investigator — Clalit Health Services; Raz Somech, MD PhD, Principal Investigator — Sheba Medical Center
Locations (4):
- Israel (4):
  - Maccabi Haifa Swimming Club, Haifa
  - Bnei Herzlyia Swimming Club, Herzlyia
  - Hod Hasharon Swimming Club, Hod HaSharon
  - Maccabim-Reut Swimming Club, Maccabim

REFERENCES:
- [Derived] Dubnov-Raz G, Rinat B, Hemila H, Choleva L, Cohen AH, Constantini NW. Vitamin D supplementation and upper respiratory tract infections in adolescent swimmers: a randomized controlled trial. Pediatr Exerc Sci. 2015 Feb;27(1):113-9. doi: 10.1123/pes.2014-0030. Epub 2014 Jul 15. PMID 25050610